CLINICAL TRIAL: NCT00841594
Title: MXQ-503 Applied To The Hand Vs. Nitroglycerin Ointment 2%, USP, Applied To The Chest: A Pharmacokinetic Comparison In Normal Subjects
Brief Title: MQX-503 Applied to the Hand Versus Nitroglycerin Ointment Applied to the Chest: A Pharmacokinetic Comparison
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MediQuest Therapeutics (Industry)
Responsible Party: Fredrick Dechow, President and CEO, MediQuest Therapeutics, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 08-001
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Raynaud's Phenomenon
Keywords: healthy volunteers
MeSH Terms: conditions — Raynaud Disease | interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): MQX-503, topical cream for nitroglycerin 0.9% vs Nitroglycerin ointment 2%, USP.
  Applied to the hand.
  Interventions: Drug: nitroglycerin 0.9 % (MXQ-503)
- 2 (Active Comparator): MQX-503, topical cream for nitroglycerin 0.9% vs Nitroglycerin ointment 2%, USP.
  Applied to the chest.
  Interventions: Drug: Nitroglycerin ointment 2%, USP

INTERVENTIONS:
Drug: nitroglycerin 0.9 % (MXQ-503) — MQX-503, topical cream for nitroglycerin 0.9% vs Nitroglycerin ointment 2%, USP.
  Arms: 1
Drug: Nitroglycerin ointment 2%, USP — MQX-503, topical cream for nitroglycerin 0.9% vs Nitroglycerin ointment 2%, USP.
  Arms: 2

SUMMARY:
The purpose of this clinical study is to compare the pharmacokinetic profiles of a topical cream formulation of 0.9% nitroglycerin, MQX 503, and Nitroglycerin Ointment 2%, USP.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age
* Subjects who do not take any prescription medication or who can safely discontinue use prior to visit 1.
* Negative pregnancy test for fertile women and agree to use effective contaception throughout the study.

Exclusion Criteria:

* Subjects who can not safely discontinue current prescription medications.
* Subjects who have a known allergy to nitroglycerin or common topical formulation ingredients.
* Subjects with an unstable medical problem.
* Subjects who, within the past three months, have had either a myocardial infarction, uncontrolled congestive heart failure, unstable angina, uncontrolled hypotension, or uncontrolled hypertension.
* Subjects who participated in a study of any investigational drug or device within four weeks prior to Visit 1.
* Subjects who have screening laboratory values which are outside the normal range and which are considered to be clinically significant to the investigator.
* Subjects who have had major abdominal, thoracic, or vascular surgery within six months of Visit 1.
* Subjects with non-epithelialized skin lesions or interfering skin conditions at time of screening in the area where either study medication is to be applied.
* Pregnant or nursing women.
* Women of childbearing potential who are unable or unwilling to comply with the contraceptive requirements during the study period.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Measurement and comparison of the levels of nitroglycerin and its dinitrate metabolites in the blood of healthy human volunteers after a single topical dose of MQX 503 and a single topical dose of Nitroglycerin Ointment 2%, USP. | 12 hours

SECONDARY OUTCOMES:
Observation for any adverse events such as headache. | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Charles River Clinical Services, Tacoma, Washington, United States